CLINICAL TRIAL: NCT02172053
Title: Effectiveness of a Resistance Training Program in the Workplace to Muscle Fatigue Control in Industrial Workers: Cluster Randomized Controlled Trial.
Brief Title: Resistance Exercise to Improve Fatigue in Workplace (REW)
Acronym: REW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosimeire Simprini Padula (Other)
Responsible Party: Sponsor-Investigator, Rosimeire Simprini Padula, PhD, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 454.709
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Fatigue; Musculoskeletal Diseases
Keywords: Workplace; Industrial workers; Resistance exercise; Fatigue; Occupational risk; Physical therapy
MeSH Terms: conditions — Fatigue; Musculoskeletal Diseases | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compensatory Workplace Exercise (CWE) (Active Comparator): Comparative Group will receive a light training protocol including warming up, stretching and resisted exercise using elastic bands.
  Interventions: Other: Compensatory Workplace Exercise (CWE) - Comparative Group
- Individual Resistance Exercise (IRE) (Experimental): Intervention group will receive training protocol including warming up, stretching a specific resistance training with increase progressive load.
  Interventions: Other: Individual Resistance Exercise (IRE) - Intervention Group

INTERVENTIONS:
Other: Compensatory Workplace Exercise (CWE) - Comparative Group — The comparative group will receive warming up and stretching and light resisted exercise with elastic bands. The exercise will realize three times per week, 20 minutes for day in total 60 minutes per week. With warming up for 5 minutes and 15 minutes of the specific training . The exercise will realize in 3 series with 10 repetitions and rest 30 seconds between series.
  Arms: Compensatory Workplace Exercise (CWE)
Other: Individual Resistance Exercise (IRE) - Intervention Group — Intervention group will receive warming up and stretching, and a specific resistance training with increase progress load. The exercise will realize three times per week, 20 minutes for day in total 60 minutes per week. With warming up and stretching for 5 minutes and 15 minutes of the specific training. The exercise will realize in 3 series with 10 repetitions and rest 30 seconds between series.
  Arms: Individual Resistance Exercise (IRE)

SUMMARY:
Studies show that exercise resistance in workplace can reduce the symptoms of induced labor, however, the effectiveness of such programs depends on the characteristics of the training fatigue. Thus, it is expected that this study the intervention group with training heavy using progressive resistance exercise protocol will be better in reducing fatigue when compare with light training group.

DETAILED DESCRIPTION:
Background: This study is randomized clinical trial with double-blinded. The aim is evaluate the effectiveness the training heavy with resistance exercise program in the muscle fatigue control. Methods: This is a randomized controlled trial by cluster, in which workers who participate in the intervention group will perform resistance exercise protocols; and workers in the comparative group held only stretching exercises and light resistance training with elastic bands. Expected results: strong evidence that fatigue reducing after ten weeks in workers and improve in others outcomes. Not found in literature studies in occupational evaluating this aspect of training.

ELIGIBILITY:
Inclusion Criteria:

* sign informed consent

Exclusion Criteria:

* restriction by the medical department.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Need for Recovery | up to 4 months
  Psychosocial risk factors and stress, resulting in work-induced fatigue, will be obtained by e Need for Recovery Scale (NFR).
Fatigue | up to 4 months
  1 RM test is the maximum amount of weight lifted once while performing a standardized exercise for muscle groups - elbow , knee and ankle flexors and extensors, trunk. A weight according to the maximum capacity is chosen. If a replay is completed, find the value of 1RM.

SECONDARY OUTCOMES:
Musculoskeletal symptoms | Outcome measures will be assessed at baseline and after 4 months.
  Musculoskeletal symptoms (pain, tingling or numbness) will be assessed using the Nordic Questionnaire for Musculoskeletal.
Level of physical activity | Outcome measures will be assessed at baseline and after 4 months.
  Questionnaire Baeck will be used to identify the level of habitual physical activity
Perceived exposure | Outcome measures will be assessed at baseline and after 4 months.
  The perception of workers risk factors that may contribute to the development of musculoskeletal complaints will be evaluated through the Job Factors Questionnaire.
Physical Fitness Assessment | Outcome measures will be assessed at baseline and after 4 months.
  The physical assessment will be consider adipometry (body fat percentage) others variables.
Productivity | Outcome measures will be assessed at baseline and after 4 months.
  Productivity is measured by a single item General Health Questionnaire and Performance at Work

CONTACTS AND LOCATIONS:
Overall Officials: Rosimeire S Padula, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Centro Universitário São Camilo, Cachoeiro de Itapemirim, Espírito Santo, Brazil

REFERENCES:
- [Derived] Santos HG, Chiavegato LD, Valentim DP, Padula RS. Effectiveness of a progressive resistance exercise program for industrial workers during breaks on perceived fatigue control: a cluster randomized controlled trial. BMC Public Health. 2020 Jun 3;20(1):849. doi: 10.1186/s12889-020-08994-x. PMID 32493267
- [Derived] Santos HG, Chiavegato LD, Valentim DP, da Silva PR, Padula RS. Resistance training program for fatigue management in the workplace: exercise protocol in a cluster randomized controlled trial. BMC Public Health. 2016 Dec 22;16(1):1218. doi: 10.1186/s12889-016-3872-5. PMID 28003034